CLINICAL TRIAL: NCT07366333
Title: Implementation of ThriveCircles for Clinician and Scientist Well-Being at CU SOM
Brief Title: ThriveCircles for Well-Being at CU SOM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Lotte Dyrbye, Senior Associate Dean for Faculty Wellbeing, Chief Well-being Officer, University of Colorado, Denver
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 262344
Record Dates: First submitted 2025-12-29; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Well-being at Work
Keywords: Clinician burnout reduction study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Thrive Circle (Experimental): Participate in small group discussions immediately
  Interventions: Behavioral: ThriveCircle Peer-Led Well-Being Groups
- Control (Delayed Intervention) (No Intervention): Wait listed control group

INTERVENTIONS:
Behavioral: ThriveCircle Peer-Led Well-Being Groups — The ThriveCircle intervention consists of peer-led small-group sessions designed to strengthen connection, reflection, and well-being among faculty. Groups of 8-10 participants meet in person six times over six months to engage in structured conversations about meaning in work, shared challenges, professional identity, and resilience, using a standardized discussion guide. Sessions include shared meals to promote community and engagement.
  Each group is self-facilitated by a faculty participant who receives brief training and a turnkey toolkit that includes facilitation guides, scheduling resources, fidelity checklists, and adaptation logs.
  Arms: Immediate Thrive Circle

SUMMARY:
This study is testing a program called ThriveCircle, which brings small groups of faculty members together to talk about their work experiences, support one another, and build a stronger sense of community. These groups meet over shared meals and use guided conversations to help reduce burnout and improve well-being among clinicians and scientists.

DETAILED DESCRIPTION:
The ThriveCircle Study is a pragmatic, hybrid Type 1 effectiveness-implementation project designed to evaluate a structured yet self-facilitated small-group program intended to improve well-being among faculty at the University of Colorado School of Medicine (CU SOM). The initiative adapts core elements from previous peer-support interventions-most notably the COMPASS model-into a format optimized for scalability, flexibility across faculty roles, and sustainable integration into institutional culture.

Study Purpose and Rationale Clinician and scientist burnout continues to rise nationally, with consequences that extend beyond individual distress to workforce instability, increased turnover intention, and patient-safety risks. Existing evidence highlights the potential of relational, community-building interventions to reduce emotional exhaustion and depersonalization and to increase professional fulfillment. However, most prior studies were conducted before 2024, in resource-intensive facilitated formats, or without examining broader outcomes such as sense of belonging, self-valuation, or imposter phenomenon.

ThriveCircle seeks to address these gaps by evaluating a contemporary, low-resource, peer-led model that emphasizes social connection, reflective dialogue, and collegial support. The program integrates commensality (shared meals), which has demonstrated additional benefit in prior studies by lowering barriers to participation and promoting trust and engagement.

Intervention Model ThriveCircle consists of six structured small-group sessions delivered over six months. Groups include approximately 8-10 faculty members and are self-facilitated by a participant who receives basic orientation and a standardized guide. The curriculum centers on meaning in work, professional identity, collegial connection, and shared challenges, with optional adaptations for scientists and for specific professional cultures. Sessions are held in person and incorporate shared meals to support accessibility and sociability.

The intervention is "light-touch," requiring minimal external facilitation, and is designed to be portable across diverse academic units. The study includes a wait-list crossover structure to ensure all participants experience the program while enabling comparative analysis of early versus delayed exposure.

Study Structure and Flow Participants complete surveys at baseline, midpoint, and endpoint to assess changes in well-being, relational factors, and other constructs relevant to burnout and professional fulfillment. Throughout the intervention period, groups maintain attendance logs and brief session check-ins documenting fidelity to core elements and any adaptations made to improve fit.

Qualitative components-including facilitator debriefs and a purposive sample of participant interviews-provide insight into mechanisms of action, contextual influences, barriers and facilitators of engagement, and perspectives on long-term sustainment.

The design acknowledges both individual-level and group-level processes. Participants are nested within groups, and analyses account for clustering and heterogeneity across departments, faculty roles, and career stages.

Implementation Evaluation To complement the assessment of effectiveness, the study incorporates a structured implementation evaluation using principles from the RE-AIM framework.

Qualitative and Mixed-Methods Components The qualitative strategy includes semi-structured interviews with facilitators and selected participants, designed to explore lived experience within circles, perceived benefits, suggestions for improvement, and contextual factors shaping group dynamics. Adaptations made during the program, team cohesion elements, perceived psychological safety, and reflections on professional meaning serve as central thematic domains. Analyses use iterative coding, triangulation, and integration with quantitative findings to enhance explanatory understanding.

Intervention Environment and Support Structure The study is situated within CU SOM's broader well-being strategy. Facilitators receive orientation, session materials, scheduling resources, and administrative support. Meal reimbursement and modest facilitator incentives support feasibility. A turnkey toolkit-including discussion guides, fidelity checklists, scheduling templates, reimbursement workflows, and adaptation logs-supports standardized yet flexible implementation.

Study staff provide ongoing communication, troubleshoot logistical issues, and monitor fidelity through routine check-ins. While groups are largely autonomous, this infrastructure promotes consistency and ensures adherence to core program components.

Data Handling and Confidentiality Practices Data collection uses secure, encrypted institutional platforms, with restricted access for authorized study personnel. Identifiers are stored separately from response data, and participant confidentiality is emphasized in both surveys and group settings. No clinical records or health information are collected. As part of institutional well-being initiatives, coded identifiers may be shared with an external survey vendor to link participation with existing biennial faculty well-being survey datasets; only de-identified data return to investigators.

Safety Considerations The intervention is non-clinical and low risk. Sessions involve reflective dialogue, which may occasionally evoke discomfort or emotional reactions. Facilitators are trained to recognize distress and direct participants to appropriate institutional resources. Adverse events-though unlikely-are documented according to institutional standards, with prompt reporting of unanticipated problems.

Participants may withdraw consent or discontinue group participation at any time. Group-level issues (e.g., persistent conflict) may prompt restructuring or, rarely, discontinuation of a circle, with continued follow-up for research purposes when appropriate.

Overall Significance The ThriveCircle Study aims to contribute rigorous, contemporary evidence on peer-led approaches to addressing burnout among faculty in academic medical centers. By pairing effectiveness testing with implementation evaluation, the project will inform scalable, sustainable strategies for promoting well-being, belonging, and retention in health sciences environments. The findings will also contribute to national conversations on how institutions can support clinicians and scientists through relational and community-based approaches rather than relying solely on individual-level interventions.

ELIGIBILITY:
Inclusion Criteria:

* Employed or affiliated faculty at CU SOM (including both CU SOM-paid and non-paid faculty)
* ≥0.5 Full-Time Equivalent (FTE) appointment
* Age 18 years or older
* Willing and able to provide informed consent
* Willing to participate in ThriveCircle group sessions (in-person, with shared meals)
* Able to communicate in English (study materials and sessions will be conducted in English)

Exclusion Criteria:

* • Faculty with <0.5 FTE appointment

  * Not affiliated with CU SOM
  * Under age 18
  * Unable or unwilling to provide informed consent
  * Unable to participate in in-person group sessions (e.g., due to geographic distance or scheduling conflicts)
  * Current participation in another well-being/job satisfaction intervention

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Maslach Burnout Inventory | From enrollment to the end of the intervention at 6 months
  Maslach Burnout Inventory - Human Services Survey for Medical Personnel (MBI-HSS MP) is a 22-item survey that covers 3 areas: Emotional Exhaustion (EE, range 0-54, higher score greater EE), Depersonalization (DP, range 0 - 30, higher score greater DP), and low sense of Personal Accomplishment (PA, range 0 -48, higher score greater PA). Each subscale includes multiple questions with frequency rating choices of Never, A few times a year or less, Once a month or less, A few times a month, Once a week, A few times a week, or Every day.

SECONDARY OUTCOMES:
Maslach Areas of Worklife Survey (AWS) - Community subscale | From enrollment to the end of the intervention at 6 months
  Maslach Areas of Worklife Survey (AWS) - Community subscale uses a 5 point Likert response format (range 1 to 5) with score computed as the average of its item responses. Higher score is favorable - meaning respondent feels well supported.
Patient Reported Outcomes Measurement Information System (PROMIS) Short Form v2.0 Social Isolation 4a scale | From enrollment to the end of the intervention at 6 months
  The PROMIS (Patient-Reported Outcomes Measurement Information System) Social Isolation Short Form v2.0 - 4a is a 4-item patient-reported outcome measure designed to assess perceptions of being excluded, detached, unknown, or disconnected from others (i.e., subjective social isolation). It is part of the NIH-supported PROMIS instrument bank for social health. Raw score range: 4 (least frequent isolation) to 20 (most frequent isolation). Scores are typically converted to a PROMIS T-score (standardized metric with mean = 50, SD = 10 in the U.S. general population) for interpretation in research and clinical contexts.
Belonging (Investigator developed) | From enrollment to end of intervention at 6 months
  Adapted from the belonging assessment used in Hunderfund et al., Sense of Belonging Among Medical Students, Residents, and Fellows: Associations with Burnout, Recruitment Retention, and Learning Environment (Acad Med, 2025). Two items capturing participants' self-reported sense of belonging within key institutional contexts (e.g., program/school and organization). The items are selected from the larger belonging assessment utilized in the referenced study to reflect core aspects of perceived inclusion, acceptance, and connectedness within the training and work environment. Ordinal Likert-type response options (e.g., 1 = Strongly disagree to 5 = Strongly agree); consistent with common belonging measures and the broader literature on belonging items. Higher scores indicate a stronger sense of belonging. Belonging has been shown to correlate with burnout outcomes, recruitment/retention indicators, and modifiable learning environment factors in medical learners.
Stanford Professional Fulfillment Index | From enrollment to end of intervention at 6 mo
  Stanford Professional Fulfillment Index (PFI) - a validated, 16-item self-report instrument designed to measure professional fulfillment (positive aspects of work) and burnout (work exhaustion and interpersonal disengagement) among physicians and other healthcare professionals. It has been widely used in well-being research and shown to be sensitive to change attributable to interventions impacting professional well-being.Professional Fulfillment (PF): 6 items assessing intrinsic positive reward from work (e.g., meaningfulness, satisfaction, sense of contribution). Work Exhaustion (WE): 4 items measuring symptoms analogous to emotional exhaustion. Interpersonal Disengagement (ID): 6 items assessing withdrawal from work relationships.Each item uses a 5-point Likert response scale (e.g., "not at all true" to "completely true" for PF items; "not at all" to "extremely" for WE and ID items). Items are scored 0-4. Scale scores are computed as the average of item scores within each subscale,
Stanford Self-Valuation Scale | From enrollment to end of intervention at 6 months
  The scale comprises 4 items, each reflecting core aspects of self-valuation including prioritization of personal well-being, learning from errors, and balancing self-care with work demands. Respondents rate each item on a 5-point Likert scale.Higher total scores indicate greater self-valuation-suggesting that participants are more likely to prioritize their own well-being, respond to challenges with growth orientation, and engage in adaptive self-care behaviors. Self-valuation has been shown to be associated with burnout and sleep-related impairment in physicians, with each point increase in self-valuation linked to significantly lower burnout scores, highlighting its potential importance as an outcome and mediator in well-being interventions.
4-item version of the Clance Imposter Phenomenon Scale | Enrollment to post intervention at 6 mo
  This abbreviated 4-item version of the Clance Impostor Phenomenon Scale was used in published research on physicians, derived from the full 20-item CIPS by selecting four items with high factor loadings relevant to impostor experiences. Participants rate 4 self-report statements capturing core impostor feelings (e.g., not internalizing success, fearing exposure as a fraud). Each item is rated on a 5-point Likert scale. Higher scores indicate greater intensity of impostor phenomenon experiences (more frequent self-doubt and fear of being found incompetent).
Self-Reported Intent to leave | Enrollment to post intervention at 6 mo
  This outcome is assessed via a single self-report survey item developed for this study to capture an individual's perceived likelihood of leaving employment with the University of Colorado School of Medicine (CU SOM) within the next two years. The item is designed to serve as a pragmatic indicator of turnover intention, a commonly reported correlate of well-being, job satisfaction, and organizational climate in healthcare workforce research.Higher scores indicate a greater self-reported likelihood of leaving CU SOM within the next two years (i.e., stronger turnover intention).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No